CLINICAL TRIAL: NCT04790422
Title: Nutrition to Relieve IBS Symptoms by Targeting the Microbiota
Acronym: NUTRIMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Collaborators: Ministery of Economic affairs (Unknown); Nexira (Industry); Wecare (Other); Roquette Freres (Industry); Ingredion Incorporated (Industry); Ingredia S.A. (Industry); Naturex (Other); Winclove Probiotics B.V. (Industry); Bioiberica (Industry); Darling Ingredients (Unknown)
Responsible Party: Principal Investigator, Diederik Esser, Project leader clinical trials, Wageningen University and Research
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NL75824.041.20
Record Dates: First submitted 2021-03-04; First posted 2021-03-10 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: gut Microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Dietary fiber 1 (Experimental)
  Interventions: Dietary Supplement: Dietary fiber supplement
- Dietary fiber 2 (Experimental)
  Interventions: Dietary Supplement: Dietary fiber supplement
- dietary fiber 3 (Experimental)
  Interventions: Dietary Supplement: Dietary fiber supplement
- caseine protein hydrolisate (Experimental)
  Interventions: Dietary Supplement: Caseine protein hydrolisate
- Maltodextrine (Placebo Comparator)
  Interventions: Dietary Supplement: Maltrodextrine

INTERVENTIONS:
Dietary Supplement: Dietary fiber supplement — Dietary fiber
  Arms: Dietary fiber 1; Dietary fiber 2; dietary fiber 3
Dietary Supplement: Caseine protein hydrolisate — Dietary supplement
  Arms: caseine protein hydrolisate
Dietary Supplement: Maltrodextrine — Placebo comparator
  Arms: Maltodextrine

SUMMARY:
Rationale: Irritable Bowel Syndrome (IBS) is functional gastrointestinal disorder that affects a large number of people. To date, no adequate treatment is available. This is partially due to the heterogeneity of the patients and the complicated pathology in which not all mechanisms are understood.

Based on results of in vitro screening within the IBSQUtrition project, we selected promising dietary supplements for validation of their potential beneficial effects on the microbiota of IBS patients.

Objective: The primary objective is to determine the bifidogenic effects of a 4-week intervention with one of four dietary supplements (Chondroitin sulfate, NOVELOSE® 3490, and Pea Fiber, and Lactium®) in IBS patients. The secondary objective is to determine the effects of the same intervention on fecal microbiota composition and SCFA concentration, IBS-related complaints, Quality of Life, and stool frequency and consistency in IBS patients.

Study design: a double-blind, randomized, placebo-controlled trial with five parallel arms. Study population: 70 adult (18-65 yrs) IBS patients Intervention: 4-week intervention period with five parallel arms: 1) Chondroitin sulfate, 2) NOVELOSE® 3490, 3) Pea Fiber, 4) Lactium®, and 5) Placebo supplement (Maltodextrin control), during which the study participants consume the respective supplement twice per day.

Main study parameters/endpoints: The main study parameter is the (relative) abundance of fecal Bifidobacterium. The secondary study parameters are fecal microbiota composition and Short-Chain Fatty Acids (SCFAs) concentration, stool frequency and consistency, IBS-related complaints, and Quality of Life (QoL).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Study participants have to invest about 7.4 hours of their time in this study mainly to complete several questionnaires (short daily questionnaire, longer questionnaires at two occasions), which is conveniently all possible from home. On two occasions they have to collect stool (transported via courier to the research facility). They have to comply to consume a commercially available supplement twice daily for four weeks. There are limited risks for the study participants.

ELIGIBILITY:
Inclusion Criteria:

* IBS patients that meet the Rome IV criteria. This will be evaluated by the medical supervisor;
* Male and female adults, aged 18-65 years;
* Having a Body Mass Index (BMI) between 18.5 and 30 kg/m2;
* Willing to keep a stable dietary pattern throughout the study;
* Having a smartphone to fill out the daily questionnaires.

Exclusion Criteria:

* Having a gastro-intestinal disease, such as celiac disease, Crohn's disease, or Ulcerative colitis;
* Having a history of intestinal surgery that might interfere with study outcomes. This does not include an appendectomy or cholecystectomy;
* Having a food allergy to milk protein or pulse protein;
* Presence of significant systemic diseases, such as diabetes mellitus, cancer, cardiovascular disease or respiratory disease;
* When applicable: currently pregnant or breastfeeding, or intending to become pregnant during the study, as this can affect stool patterns and wellbeing;
* Use of antibiotic treatment less than 3 months before start of the study and no use of antibiotics during the study;
* Use of prebiotics and/or probiotics (should be stopped 4 weeks before the start of the study) and infrequent use of other (fiber) supplements. Some supplements are allowed, but intake should be kept stable during the whole study period (Supplements will be judged by the medical supervisor MD Ben Witteman);
* Currently following a FODMAP-restricted diet;
* Use of medication that can interfere with the study outcomes, including anxiolytics, proton pump inhibitors, laxatives (Over-the-counter laxatives are allowed, but intake should be either stopped before the start of the study or kept stable during the complete study period), and codeine, as judged by the medical supervisor MD Ben Witteman;
* Participation in another clinical trial at the same time;
* Student or employee working at Food, Health and Consumer Research from Wageningen Food and Biobased Research;
* Alcohol intake ≥ 2 (women) or ≥ 4 (men) glasses of alcoholic beverages per day;
* Abuse of illicit drugs;
* Being incapacitated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Abundance of feceal Bifidobacterium | Change after the intervention of 4 weeks
  Measured in fecal samples using 16S rRNA gene-based approaches

SECONDARY OUTCOMES:
fecal microbiota composition | Change after the intervention of 4 weeks
  Measured in fecal samples using 16S rRNA gene-based approaches
fecal microbiota metabolite levels | Change after the intervention of 4 weeks
  Measured in the fecal samples using HPLC
Stool frequency | daily during 4 weeks
  Questions regarding how often participants defecate
Stool consistency | daily during 4 weeks
  Using the validated Bristol stool chart
gastro-intestinal complaints | daily during 4 weeks
  Measured with a visual analog scale
Irritable Bowel Syndrome severity | 4 weeks
  measured using the validated IBS-SSS questionnaire
Irritable Bowel Syndrome related quality of life | 4 weeks
  measured using the validated IBS-QoL questionnaire
mental wellbeing | 4 weeks
  measuring using the validated hospital anxiety and despression score (HADS) questionnaire
dietary intake | 4 weeks
  Measured via a validated food frequency questionnaire (FFQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No